CLINICAL TRIAL: NCT03324464
Title: Central Executive Training for ADHD: Efficacy Trial
Brief Title: Central Executive Training (CET) for ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Kofler, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH115048 (NIH)
Record Dates: First submitted 2017-10-09; First posted 2017-10-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CET-Working Memory (WM) (Experimental): Central Executive Training: Working Memory
  Interventions: Behavioral: Central Executive Training: Working Memory
- CET-Behavioral Inhibition (BI) (Active Comparator): Central Executive Training: Inhibitory Control
  Interventions: Behavioral: Central Executive Training: Inhibitory Control

INTERVENTIONS:
Behavioral: Central Executive Training: Working Memory — Computerized working memory training
  Arms: CET-Working Memory (WM)
Behavioral: Central Executive Training: Inhibitory Control — Computerized inhibitory control training
  Arms: CET-Behavioral Inhibition (BI)

SUMMARY:
The goal of the current project is to assess the efficacy of Central Executive Training (CET) for youth with ADHD. CET is a new, computerized training intervention that targets specific components of the working memory system. Two versions of CET were developed as part of our R34, each targeting a different combinations of executive functions. The final CET protocol reflects the contributions and feedback of a diverse group of caregivers, children with ADHD, and recognized experts in human cognition, ADHD treatment research, randomized control trial (RCT) intervention design methods, serious game theory and task design, cognitive training, and the role of executive dysfunction in ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-12 with principal ADHD diagnoses (via Kiddie Schedule for Affective Disorders semi-structured clinical interviewing (K-SADS)
* Parent AND teacher ratings in clinical/borderline range based on age and gender on ADHD-RS-5 or BASC-3 Attention Problems/Hyperactivity subscales
* Below average or lower working memory on at least one pre-treatment WM test. All ADHD presentations will be eligible.

Exclusion Criteria:

* gross neurological, sensory, or motor impairment
* history of seizure disorder, psychosis, bipolar, or severe dysregulation disorders that may interfere with study participation (substance use, disruptive mood dysregulation, intermittent explosive, reactive attachment)
* intellectual disability or Wechsler Intelligence Scale for Children (WISC-V) short-form intelligence quotient (FSIQ) < 78 (1.5 standard deviations (SD) below mean)
* conditions requiring acute intervention, e.g., active suicidality
* non-English speaking child or parent.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms | Immediate post-treatment (within 2 weeks of final treatment session)
  Average of T-scores on parent-report ADHD symptoms questionnaires (Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-5) Inattention and Hyperactivity subscales, Behavioral Assessment System for Children (BASC-3) Inattention and Hyperactivity subscales)

SECONDARY OUTCOMES:
Working Memory | Immediate post-treatment (within 2 weeks of final treatment session)
  Average of stimuli correct per trial on the Rapport phonological and visuospatial working memory tests
Inhibitory control | Immediate post-treatment (within 2 weeks of final treatment session)
  Average of performance on the stop-signal (stop-signal delay metric) and go/no-go tests (commission errors)
Actigraph-measured hyperactivity during working memory testing | Immediate post-treatment (within 2 weeks of final treatment session)
  Proportional integrating measure (PIM) units from autographs worn on non dominant wrist, left ankle, and right ankle during Rapport working memory tests. PIM units from each actigraph will be aggregated by summing them to create a Total Hyperactivity Score.
Actigraph-measured hyperactivity during baseline | Immediate post-treatment (within 2 weeks of final treatment session)
  Proportional integrating measure (PIM) units from autographs worn on non dominant wrist, left ankle, and right ankle. During beginning and end of session baseline painting tasks (described in Rapport et al., 2009). PIM units from each actigraph will be aggregated by summing them to create a Total Hyperactivity Score.

OTHER OUTCOMES:
NIH List Sorting | Follow-up testing: 2-4 months after the post-treatment evaluation (variable time frame to account for school breaks)
  Standard scores on NIH List Sorting test
Teacher-reported ADHD symptoms | Immediate post-treatment (within 2 weeks of final treatment session)
  Average of T-scores on teacher-report ADHD symptoms questionnaires (ADHD-5 Inattention and Hyperactivity subscales, BASC-3 Inattention and Hyperactivity subscales)
Academic performance rating scale (APRS) | Immediate post-treatment (within 2 weeks of final treatment session)
  Total score (T-score) for academic performance (teacher ratings)
Children's Organizational Skills Scale (COSS) Parent Report | Immediate post-treatment (within 2 weeks of final treatment session)
  Parent-reported total organizational problems (T-score)
Children's Organizational Skills Scale (COSS) Teacher Report | Immediate post-treatment (within 2 weeks of final treatment session)
  Teacher-reported total organizational problems (T-score)
Social Skills: Parent Report | Immediate post-treatment (within 2 weeks of final treatment session)
  Parent-reported total score (standard score) on Social Skills Improvement System (SSIS)
Social Skills: Teacher Report | Immediate post-treatment (within 2 weeks of final treatment session)
  Teacher-reported total score (standard score) on Social Skills Improvement System (SSIS)
Parent-child relationship quality | Immediate post-treatment (within 2 weeks of final treatment session)
  Parent-reported total score (T-score) on Parent Relationship Questionnaire (PRQ)
Kaufman Test of Educational Achievement Third Edition (KTEA-3) Reading Comprehension | Follow-up testing: 2-4 months after the post-treatment evaluation (variable time frame to account for school breaks)
  Standard score on KTEA-3 Reading Comprehension subtest
Kaufman Test of Educational Achievement Third Edition (KTEA-3) Listening Comprehension | Follow-up testing: 2-4 months after the post-treatment evaluation (variable time frame to account for school breaks)
  Standard score on KTEA-3 Listening Comprehension subtest
Kaufman Test of Educational Achievement Third Edition (KTEA-3) Reading Fluency | Follow-up testing: 2-4 months after the post-treatment evaluation (variable time frame to account for school breaks)
  Standard score on KTEA-3 Reading Fluency subtest
Kaufman Test of Educational Achievement Third Edition (KTEA-3) Math Fluency | Follow-up testing: 2-4 months after the post-treatment evaluation (variable time frame to account for school breaks)
  Standard score on KTEA-3 Math Fluency subtest

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Groves NB, Chan ESM, Marsh CL, Gaye F, Jaisle EM, Kofler MJ. Does central executive training and/or inhibitory control training improve emotion regulation for children with attention-deficit/hyperactivity disorder? A randomized controlled trial. Front Psychiatry. 2022 Dec 6;13:1034722. doi: 10.3389/fpsyt.2022.1034722. eCollection 2022. PMID 36561637